CLINICAL TRIAL: NCT00025402
Title: Randomized Multicenter Treatment Optimization Study In Chronic Myeloid Leukemia (CML) Interferon-a Vs. Allogeneic Stem Cell Transplantation Vs. High-Dose Chemotherapy Followed By Autografting And Interferon-a Maintainance In Early Chronic Phase
Brief Title: Chemotherapy and Biological Therapy With or Without Bone Marrow or Peripheral Stem Cell Transplant in Treating Patients With Chronic Myelogenous Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: III. Medizinische Klinik Mannheim (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068957; III-MK-CML-3A; EU-20118
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-07

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; Philadelphia chromosome negative chronic myelogenous leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Filgrastim; Interferon-alpha; Busulfan; Cyclophosphamide; Cytarabine; Etoposide; Hydroxyurea; Idarubicin; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Drug: hydroxyurea
Drug: idarubicin
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy, such as hydroxyurea, cytarabine, idarubicin, and etoposide before a donor bone marrow transplant or stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Interferon alfa may interfere with the growth of cancer cells and slow the growth of cancer. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known whether chemotherapy is more effective with or without interferon alfa and/or bone marrow or stem cell transplant in treating patients with chronic myelogenous leukemia.

PURPOSE: This randomized phase III trial is studying chemotherapy and biological therapy to see how well it works compared with chemotherapy, biological therapy, and donor bone marrow transplant or autologous stem cell transplant in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival in patients with chronic myelogenous leukemia in early chronic phase treated with allogeneic bone marrow transplantation vs drug treatment with or without autologous peripheral blood stem cell transplantation.
* Compare survival of patients with late-phase disease treated with high-dose cytarabine vs low-dose cytarabine followed by autografting and interferon alfa maintenance.
* Compare survival of patients not responding cytogenetically to treatment with continued interferon alfa vs hydroxyurea.
* Determine frequency, time-point, and duration of hematological and cytogenetic remissions and of Philadelphia chromosome-negative and/or BCR-ABL-positive cells on the various treatments.
* Correlate the quality of hematological and cytogenetic remissions with survival time in patients treated with these regimens.
* Compare the course of the terminal phase in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Determine the effect of prognostic criteria and normal or subnormal WBC on chronic phase duration and survival time in patients treated with these regimens.
* Compare the effect of early vs late high-dose therapy plus autografting on feasibility, toxicity, and survival times in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to eligibility for transplantation (yes vs no).

All patients undergo cytoreduction comprising hydroxyurea (HU) IV daily.

Patients who are ineligible for or refuse transplantation are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive interferon alfa (IFN) subcutaneously (SC) daily. After 2 weeks of IFN therapy, patients also receive low-dose cytarabine (ARA-C) SC once daily for 10-15 days each month. Patients who do not achieve cytogenetic remission within 12 months continue to receive HU.
* Arm II: Patients receive IFN SC daily. After 2 weeks of IFN therapy, patients also receive low-dose ARA-C SC daily for 10-15 days each month. Patients who do not achieve cytogenetic remission within 12 months continue to receive IFN therapy SC daily.

Patients who are eligible for transplantation with a related donor undergo allogeneic bone marrow transplantation. Patients may receive HU or IFN prior to transplantation. Patients may also receive oral high-dose busulfan daily for 4 days with or without cyclophosphamide or cyclophosphamide with total body irradiation.

Patients who are eligible for transplantation but do not have a related donor undergo peripheral blood stem cell (PBSC) harvest and are randomized to 1 of 2 treatment arms.

* Arm III: Patients receive IFN and low-dose ARA-C as in arm I. Patients who accelerate on treatment may undergo autologous PBSC transplantation.
* Arm IV: Patients receive idarubicin IV, ARA-C IV over 2 hours, and etoposide IV on days 1-3. Patients then undergo leukapheresis. Beginning on day 8, patients receive filgrastim (G-CSF) SC daily until end of leukapheresis. Patients then receive oral high-dose busulfan daily for 4 consecutive days. The following day, patients undergo reinfusion of autologous PBSC. After blood count recovery, patients receive maintenance IFN 3 times weekly for 8 weeks and then daily.

Patients are followed every 3 months for 3 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia in chronic phase

  * Previously untreated
* Patients negative for Philadelphia chromosome and BCR-ABL translocation must fulfill at least 1 of the following criteria:

  * Impaired health status with reduced exercise tolerance
  * Spleen-related symptoms in cases of splenomegaly
  * Weight loss greater than 10% in 6 months
  * Fever greater than 38.5 degrees C on 5 consecutive days
  * Clinically relevant bone pain
  * Leukocytosis greater than 5,000/mm^3
  * Thrombocytosis greater than 100,000/mm^3

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent malignancy that is likely to require treatment during study or that is likely to reduce life expectancy
* No severe concurrent disease or other cause that would preclude study
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1997-07

PRIMARY OUTCOMES:
Survival
Frequency, time-point, and duration of hematologic and cytogenetic remissions and of Philadelphia chromosome-negative and/or BCL-ABL-positive cells
Correlation of quality of hematological and cytogenetic remission with survival time
Course of the terminal phase
Toxicity
Effect of prognostic criteria and normal or subnormal WBC on chronic phase duration and survival time
Effect of early vs late high-dose therapy and autografting on feasibility, toxicity and survival times

CONTACTS AND LOCATIONS:
Overall Officials: Ruediger Hehlmann, MD, Study Chair — III. Medizinische Klinik Mannheim
Locations (187):
- Masaryk University Hospital, Brno, Czechia
- Germany (166):
  - Haematologisch Onkologische Praxis, Aachen
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Urologische Klinik - Universitaetsklinikum Aachen, Aachen
  - Kreiskrankenhaus, Aalen
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - II. Medizinische Klinik, Aschaffenburg
  - Haematologische Praxis, Augsburg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus, Bad Hersfeld
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - St. Hedwig Kranken Haus, Berlin
  - Tumorzentrum Berlin-Moabit, Berlin
  - Wenckebach - Krankenhaus, Berlin
  - Helios Klinikum Berlin, Berlin
  - Haematologisch-Onkologische Schwerpunktpraxis, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Onkolog - Haematolog Schwerpunktpraxis, Berlin
  - Krankenhaus Neukoelln, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Kinderklinik der Freier Universitaet Berlin, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Franziskus Hospital, Bietigheim
  - Krankenhaus Bietigheim, Bietigheim
  - Europahochhaus, Bochum
  - Universitaetsklinikum Bonn, Bonn
  - Medizinische Poliklinik, Bonn
  - Marienhospital Bottrop gGmbH, Bottrop
  - Kreiskrankenhaus Boeblingen, Böblingen
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - St. Joseph Hospital, Bremerhaven
  - Zentralkrankenhaus, Bremerhaven
  - Medizinische Klinik Am Lukas - Krankenhaus, Bünde
  - Klinikum Coburg, Coburg
  - Praxis Gemeinschaft, Cologne
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Onkologische Schwerpunktpraxis, Cottbus
  - Stadt. KH Dresden - Neustadt, Dresden
  - Medizinische Klinik I, Dresden
  - Michael Schaefers und Partner, Duisburg
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Krankenhaus Dueren, Düren
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Hans - Susemihl - Krankenhaus, Emden
  - Internistiche Praxis, Erfurt
  - Klinikum Erfurt, Erfurt
  - Praxis DR. J. Weniger, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - Medizinische Klinik III - Universitaetsklinikum Erlangen, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Malteser Krankenhaus, Flensburg
  - Onkolog Gemeinschaftspraxis, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - II Medizinische Klinik - Klinikum Fuerth, Fürth
  - Kreiskrankenhaus Fuessen, Füssen
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Klinik und Poliklinik fuer Urologie und Kinderurologie, Giessen
  - DR Herbert - Nieper Krankenhaus Goslar, Goslar
  - Klinik fuer Radioonkologie und Strahlentherapie, Göppingen
  - Universitaetsklinikum Goettingen, Göttingen
  - Allgemeines Krankenhaus Hagen, Hagen
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Allgemeines Krankenhaus Altona, Hamburg
  - Hermann - Holthusen Institute for Radiotherapy, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Onkologischer Schwerpunkt Lerchenfeld, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Haematologie Und Internistische Onkologie, Hanau
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Klinikum Herford, Herford
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Praxis am Evangelischen Krankenhaus Bethanien, Iserlohn
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Gemeinschaftspraxis Brunoehler, Karlsruhe
  - St. Vincentius-Kliniken, Karlsruhe
  - Diakonissen - Krankenhaus, Karlsruhe-Rueppur
  - Klinikum Kassel, Kassel
  - Klinikum Kempten Oberallgaeu, Kempten
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinik Konstanz, Konstanz
  - Haematologische / Onkologische Schwerpunktpraxis, Krefeld
  - Klinikum Krefeld GmbH, Krefeld
  - Vinzentiuskrankenhaus, Landau
  - Caritas - Krakenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Klinikum Lippe - Lemgo, Lemgo
  - Luisenkrankenhaus, Lindenfels
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - St Marienkrankenhaus, Ludwigshafen, Rhein
  - Praxis Fuer Haematologie/Onkologie, Lübeck
  - Onkologische Schwerpunktpraxis Lueneburg, Lüneburg
  - Gemeinschaftspraxis, Mannheim
  - III Medizinische Klinik Mannheim, Mannheim
  - Philipps-Universitaet Marburg Klinikum, Marburg
  - Kreiskrankenhaus Mellrichstadt, Mellrichstad
  - Klinikum Minden, Minden
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Gemeinschaftspraxis, Munich
  - Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Medizinische Kl. Klinikum Innenstadt Universitaet Muenchen, Munich
  - Praxis fuer Innere Medizin und Haematologie, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Krankenhaus Muenchen Neuperlach, Munich
  - Universitaets - Kinderpoliklinik, München
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Ruppiner Klinikum GMBH, Neuruppin
  - Gemeinschaftspraxis, Niddatel-IIbenstadt
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Gemeinschaftspraxis, Nuremberg
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum Nuernberg - Klinikum Sued, Nuremberg
  - Hematologische Praxis, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Paracelsus - Klinik Osnabrueck, Osnabrück
  - Staedtisches Krankenhaus, Pforzheim
  - Kreiskrankenhaus Radebeul, Radebeul
  - St. Elisabeth Krankenhaus, Ravensburg
  - Prosper-Hospital Recklinghausen, Recklinghausen
  - Hematologische Onkologische Praxis, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Klinikum Remscheid GmbH, Remscheid
  - Jakobi Krankenhaus, Rheine
  - Caritasklinik St. Theresia, Saarbrücken
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - Saechsische Schweiz Klinik, Sebnitz
  - Staedt Krankenhaus, Sebnitz
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Kreiskrankenhaus Siegen, Siegen
  - Klinikum Der Hansestadt Stralsund - Klin. West, Stralsund
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Trier
  - Praxis Fuer Internistische Haematologie / Onkologie, Troisdorf
  - Schwerpunktpraxis für Rheumatologie und Haematologie/Internistische Onkologie, Tübingen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Bundeswehr Krakenhaus, Ulm
  - Universitaetsklinikum Ulm, Ulm
  - St. Irmgardis Krankenhaus, Viersen-Suechteln
  - Klinikum Der Stadt Villingen - Schwenningen, Villingen-Schwenningen
  - Krankenhaus St. Michael, Voeklingen
  - Kreiskrankenhaus, Waldroel
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
  - St. Willehad Hospital, Wilhelmshaven
  - Praxis Fuer Haemotologie Und Internistischer Onkologie, Wuppertal
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Kliniken St. Antonius, Wuppertal
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Silesian Medical Academy, Katowice
- Hospital Universitario Virgen de la Victoria, Málaga, Spain
- Switzerland (17):
  - Kantonspital Aarau, Aarau
  - Facharzt FMH Fuer Innere Medizin and Oncology, Baar
  - Basel
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Facharzt Fuer Onkologie-Hematologie, Bern
  - Inselspital Bern, Bern
  - Inneremedizin FMH, Breitenbach
  - Bezirksspital Dornach, Dornach
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - FMH f. Innere Medizin and Hematologie, Gross Höchstetten
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Luzerne, Luzerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Institut Central des Hopitaux Valaisans, Sion
  - Klinik Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich